CLINICAL TRIAL: NCT00691418
Title: DHA Administration and Length of Gestation: a Feasibility Study
Brief Title: Docosahexaenoic Acid (DHA) Administration and Length of Gestation: a Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decision made not to proceed -- no subjects were ever enrolled
Sponsor: Kaiser Permanente (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KP-Martek01
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Premature Birth
Keywords: perinatal; premature; pregnancy; gestation
MeSH Terms: conditions — Premature Birth | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 600 mg per day of docosahexaenoic acid (DHA)
  Interventions: Dietary Supplement: docosahexaenoic acid (DHA)
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: docosahexaenoic acid (DHA) — 600 mg per day of docosahexaenoic acid (DHA) starting at 22-24 weeks gestation until delivery.
  Other Names: omega fatty acid
  Arms: 1
Dietary Supplement: placebo — placebo once per day starting at 22-24 weeks gestation until delivery.
  Arms: 2

SUMMARY:
This is a feasibility study to determine if it will be possible to conduct a larger study of the effect of docosahexaenoic acid (DHA), an omega fatty acid, on increased length of gestation among women who have had a previous preterm delivery.

DETAILED DESCRIPTION:
We propose to conduct an 18-month feasibility study to determine (a) how many women we could approach during a 4-month period, (b) how many of these women would be eligible for a future RCT, (c) how many would consent to participate in the RCT, and (d) how many would be subsequently rendered ineligible due to poor compliance. Women enrolled during the 4-month recruitment period would be followed until 1 month after delivery using telephone contact (for assessing compliance) and scanning of KPMCP electronic databases (for quantifying outcomes). We hope to enroll 50 to 75 women during our fixed time (4 months) recruitment period. Half of these 50-75 women would receive DHA; half would receive placebo.

We will identify potential subjects based on their response to the Preterm Birth Prevention Program questionnaire (a screening instrument administered by the Regional Perinatal Service Center [RPSC] to all women in the KPMCP entering prenatal care). Eligible women are those pregnant women entering prenatal care who, based on their response to the abovementioned RPSC questionnaire, are identified as having had a previous preterm delivery (delivery prior to 37 completed weeks of gestation).

Results of this study will (a) permit us to determine whether an RCT is feasible at a reasonable cost, and (b) assuming the answer to (a) is positive, it would then be possible for us to design an RCT that could address our primary study question.

ELIGIBILITY:
Inclusion Criteria:

* Previous preterm delivery (delivery prior to 37 completed weeks of gestation)

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Is daily intake of 600 mg per day of docosahexaenoic acid (DHA), a long-chain polyunsaturated fatty acid, beginning at 22-24 weeks gestation, associated with increased length of gestation among women who have had a previous preterm delivery? | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Escobar, MD, Principal Investigator — Kaiser Permanente